CLINICAL TRIAL: NCT00431964
Title: Multi-center, Multi-national, Randomized, Placebo-Controlled Trial of Azithromycin in Subjects With Cystic Fibrosis 6-18 Years Old, Culture Negative for Pseudomonas Aeruginosa
Brief Title: Effect of Azithromycin on Lung Function in 6-18 Year-olds With Cystic Fibrosis (CF) Not Infected With P. Aeruginosa
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CF Therapeutics Development Network Coordinating Center (Network)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AZ0004
Record Dates: First submitted 2007-02-02; First posted 2007-02-06 (Estimated); Results first posted 2015-08-19 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-07

CONDITIONS: Cystic Fibrosis
Keywords: azithromycin, Zithromax
MeSH Terms: conditions — Cystic Fibrosis | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active (Active Comparator): azithromycin 250 mg tablets
  Interventions: Drug: azithromycin 250 mg tablets
- Placebo (Placebo Comparator): placebo tablets (matched to active drug in appearance)
  Interventions: Drug: placebo tablets

INTERVENTIONS:
Drug: azithromycin 250 mg tablets — * One (1) tablet three times weekly for patients who weigh 40-79 lbs
  * Two (2) tablets three times weekly for patients who weigh greater than or equal to 80 lbs
  Other Names: Zithromax
  Arms: Active
Drug: placebo tablets — * One (1) tablet three times weekly for patients who weigh 40-79 lbs
  * Two (2) tablets three times weekly for patients who weigh greater than or equal to 80 lbs
  Other Names: inactive pill
  Arms: Placebo

SUMMARY:
This is a study to examine the safety, effect on lung function, and frequency of symptoms relating to cystic fibrosis during 24 weeks of treatment with the antibiotic azithromycin in 6-18 year-olds with CF who are not infected with Pseudomonas aeruginosa.

DETAILED DESCRIPTION:
Azithromycin is an antibiotic that has been shown to improve lung function in patients with cystic fibrosis (CF) whose lungs are infected with a bacterium called Pseudomonas aeruginosa. Scientists are not sure how azithromycin works in cystic fibrosis. It does not appear to work by killing the bacteria Pseudomonas aeruginosa, but it may make these bacteria and other bacteria less damaging to the lungs by reducing their ability to attach to the lining of the lung, or by reducing the bacteria's ability to make substances that damage the lungs of patients with cystic fibrosis. Azithromycin may also work directly on the cells in the lungs to improve lung function. This could occur by reducing inflammation (swelling) in the lungs, and/or making the mucus less sticky, or by affecting the salt channel that doesn't function correctly in CF. If azithromycin works in one or more of these ways; it may also be effective in improving lung function in cystic fibrosis patients who are not infected with Pseudomonas aeruginosa.

We are conducting this research study to examine the safety, effect on lung function and frequency of symptoms relating to cystic fibrosis during 24 weeks of treatment with the antibiotic azithromycin. This study is designed to determine if patients with cystic fibrosis whose lungs are not infected with the bacteria Pseudomonas aeruginosa will benefit from 24 weeks of treatment with the antibiotic azithromycin. Benefit will be determined as having better pulmonary function tests and getting sick less often compared to a placebo (sugar pill). This study is also designed to determine if azithromycin is safe when administered for 24 weeks to cystic fibrosis patients not infected with Pseudomonas aeruginosa. By doing this study, we hope to learn more about CF and improve the way in which we treat it.

Comparison: Three times weekly azithromycin tablets added to standard care, compared to three times weekly placebo tablets added to standard care.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 6-18 years of age at enrollment
* Confirmed diagnosis of CF
* Written informed consent (and assent when applicable)
* Clinically stable at enrollment as assessed by the site investigator
* FEV1 % predicted > 50%
* Ability to comply with medication use, study visits, and study procedures
* Ability to swallow a 250 mg tablet

Exclusion Criteria:

* Weight less than 18.0 kg
* Respiratory culture positive for P. aeruginosa, NTM, or B. cepacia complex within 1 year or at screening, or AFB positive at screening
* Allergy to macrolide antibiotics
* Use of macrolide antibiotics (e.g., azithromycin, clarithromycin) within 60 days of screening
* Use of systemic corticosteroids or intravenous or oral antibiotics within 14 days of screening
* Initiation of high dose ibuprofen, Pulmozyme®, hypertonic saline or aerosolized antibiotics within 30 days of screening
* Chronic therapy with drugs known to have rare but serious interactions with azithromycin: amiodarone, digoxin, disopyramide, lovastatin, pimozide, rifabutin, and nelfinavir
* Investigational drug use within 30 days of screening
* Laboratory abnormalities (creatinine, liver function or neutropenia) at screening and confirmed at follow-up testing prior to randomization
* History of biliary cirrhosis, portal hypertension, or splenomegaly, or splenomegaly on physical exam
* History of ventricular arrhythmia
* Other major organ dysfunction, excluding pancreatic dysfunction
* History of lung transplantation or currently on lung transplant list
* Relative decrease in FEV1 % predicted ≥ 20% between the screening and enrollment visit
* Positive serum pregnancy test at screening
* Pregnant, breastfeeding, or if post-menarche female, unwilling to practice birth control during participation in the study
* History of alcohol, illicit drug or medication abuse within 1 year of screening in the judgment of the site investigator
* Presence of a condition or abnormality that in the opinion of the site investigator would compromise the safety of the subject or the quality of the data

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 263 (Actual)
Dates: Start 2007-02; Primary Completion 2009-07 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Saiman, MD, MPH, Principal Investigator — Columbia University; Michael Anstead, MD, Principal Investigator — University of Kentucky; Felix Ratjen, MD, Principal Investigator — The Hospital for Sick Children, Toronto, Ontario; Larry Lands, MD, Principal Investigator — Montreal Children's Hospital of the MUHC
Locations (40):
- United States (31):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Emory University, Atlanta, Georgia
  - Children's Memorial Hospital, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Kentucky, Lexington, Kentucky
  - Children's Hospital Boston, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - Washington University, St Louis, Missouri
  - University of Nebraska Medical Center - Pediatric Pulmonary, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Columbia University, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - New York Medical College, Valhalla, New York
  - UNC Chapel Hill, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pulmonary Medicine, Allergy & Immunology, Pittsburgh, Pennsylvania
  - East Tennessee Children's Hospital, Pediatric Pulmonary & Respiratory Care, Knoxville, Tennessee
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - University of Utah Pediatric Pulmonology, Salt Lake City, Utah
  - Vermont Children's Hospital, Burlington, Vermont
  - University of Virginia at Charlottesville Children's Hospital, Charlottesville, Virginia
  - West Virginia University, Morgantown, West Virginia
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Canada (9):
  - Alberta Children's Hospital, Calgary, Alberta
  - BC Children's Hospital, Vancouver, British Columbia
  - Janeway Children's Health & Rehabilitation Hospital, St. John's, Newfoundland and Labrador
  - McMaster Health Sciences Centre, Hamilton, Ontario
  - Bryan Lyttle, MD, Private Practice, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - CSSS de Chicoutimi, Chicoutimi, Quebec
  - Montreal Children's Hospital, Montreal, Quebec

REFERENCES:
- [Result] Saiman L, Anstead M, Mayer-Hamblett N, Lands LC, Kloster M, Hocevar-Trnka J, Goss CH, Rose LM, Burns JL, Marshall BC, Ratjen F; AZ0004 Azithromycin Study Group. Effect of azithromycin on pulmonary function in patients with cystic fibrosis uninfected with Pseudomonas aeruginosa: a randomized controlled trial. JAMA. 2010 May 5;303(17):1707-15. doi: 10.1001/jama.2010.563. PMID 20442386
- [Derived] Ratjen F, Saiman L, Mayer-Hamblett N, Lands LC, Kloster M, Thompson V, Emmett P, Marshall B, Accurso F, Sagel S, Anstead M. Effect of azithromycin on systemic markers of inflammation in patients with cystic fibrosis uninfected with Pseudomonas aeruginosa. Chest. 2012 Nov;142(5):1259-1266. doi: 10.1378/chest.12-0628. PMID 22595153

RESULTS

PARTICIPANT FLOW:
Groups:
- Active: azithromycin 250 mg tablets
  azithromycin 250 mg tablets: *One (1) tablet three times weekly for patients who weigh 40-79 lbs
  *Two (2) tablets three times weekly for patients who weigh greater than or equal to 80 lbs
- Placebo: placebo tablets (matched to active drug in appearance)
  placebo tablets: *One (1) tablet three times weekly for patients who weigh 40-79 lbs
  *Two (2) tablets three times weekly for patients who weigh greater than or equal to 80 lbs
Period: Overall Study
Arm/Group | Active | Placebo
Started | 131 | 132
Randomized/Received Drug | 131 | 129
Did Not Receive Drug | 0 | 3
Withdrew From Study | 6 | 5
Completed | 125 | 124
Not Completed | 6 | 8
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 1 | 2
Not completed — Physician Decision | 2 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Parental Consent Withdrawn | 0 | 2
Not completed — Due to Unstable Health | 0 | 1

BASELINE CHARACTERISTICS:
Population: 3 participants in the Placebo arm were randomized but did not receive drug due to withdrawal of consent and unstable health.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Placebo | Total
Number analyzed (Participants) | 131 | 129 | 260
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 131 | 129 | 260
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.7 (3.25) | 10.6 (3.10) | 10.7 (3.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 59 | 113
  Male | 77 | 70 | 147

OUTCOME MEASURES:

1. Primary Outcome: Change in FEV1 From Baseline to End of Treatment at Day 168
Time Frame: change from baseline to day 168
Population: Modified intent to treat (randomized and at least one dose of study drug).
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Active | Placebo
Number analyzed (Participants) | 131 | 129
liters | 0.08 (0.25) | 0.06 (0.28)

ADVERSE EVENTS:
Time Frame: Randomization through Day 168
Arm/Group | Active | Placebo
Serious Adverse Events (participants affected / at risk) | 12/131 | 14/129
Other Adverse Events (participants affected / at risk) | 121/131 | 128/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=131) | Placebo (N=129)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1)
Exercise tolerance decreased (General disorders) | 0 (0) | 1 (1)
Implant site pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Burkholderia cepacia infection (Infections and infestations) | 1 (1) | 0 (0)
Pseudomonas infection (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Pulmonary function test decreased (Investigations) | 1 (1) | 2 (2)
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Gastrostomy tube insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Oesophagogastric fundoplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Sinus operation (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=131) | Placebo (N=129)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 9 (11)
Abdominal pain (Gastrointestinal disorders) | 11 (11) | 11 (11)
Abdominal pain upper (Gastrointestinal disorders) | 16 (23) | 20 (37)
Constipation (Gastrointestinal disorders) | 8 (10) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 11 (12)
Nausea (Gastrointestinal disorders) | 11 (15) | 12 (15)
Vomiting (Gastrointestinal disorders) | 21 (29) | 31 (40)
Fatigue (General disorders) | 9 (9) | 13 (14)
Pain (General disorders) | 0 (0) | 7 (7)
Pyrexia (General disorders) | 29 (31) | 41 (54)
Pseudomonas infection (Infections and infestations) | 9 (9) | 15 (15)
Pulmonary function test decreased (Investigations) | 8 (9) | 15 (16)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 9 (9)
Headache (Nervous system disorders) | 30 (53) | 40 (84)
Cough (Respiratory, thoracic and mediastinal disorders) | 63 (118) | 91 (172)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (12) | 9 (10)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 45 (63) | 42 (64)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 29 (40) | 43 (64)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 24 (25)
Rales (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 25 (37) | 36 (62)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 9 (10)
Rash (Skin and subcutaneous tissue disorders) | 9 (12) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No